CLINICAL TRIAL: NCT03444740
Title: Do Women Seeking Medical Assistance for Lower Urinary Tract Symptoms Have a High Prevalence of Adjustment Disorder?A Questionnaire Based Study
Brief Title: Lower Urinary Tract Symptoms in Women and Adjustment Disorder
Acronym: LUTS and AD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Basel Women's University Hospital (Other)
Responsible Party: Principal Investigator, Tilemachos Kavvadias, MD, Basel Women's University Hospital
Other Study IDs: LUTS and AD
Record Dates: First submitted 2018-02-19; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Lower Urinary Tract Symptoms; Adjustment Disorders
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Adjustment Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ICIQ-FLUTS, ADMN-20 — Questionnaire

SUMMARY:
Our hypothesis that the prevalence of AD in uro-gynecologic patients with LUTS who are seeking medical help for their condition is higher than that of the general population (indicated by high scores at the ADNM-20; score above 48). Taking into consideration that affective disorders, anxiety and depression among patients with LUTS present with a prevalence of 17-23% [20] as well as through long personal experience, we hypothesize that the prevalence of AD in this group is 20%.

ELIGIBILITY:
Inclusion Criteria:

* Female patients seeking medical help for lower urinary tract symptoms
* German speaking

Exclusion Criteria:

* Pelvic floor Prolapse symptoms or Stage III or more by medical examination
* Inability to understand the purpose of the study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All eligible female patients at first time visits or follow-up visits who present to the uro-gynecology department of the University Hospital of Basel with LUTS (such as incontinence, OAB or recurrent UTIs) will be asked to participate in the study. After counseling and agreement the patients will be asked to sign the informed consent
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of adjustment disorders among women with lower urinyry tract symptoms | 9 Months

SECONDARY OUTCOMES:
Correlation between ICIQ-FLUTS and ADNM-20 scores | 9 Months

IPD SHARING:
Plan to Share IPD: Undecided